CLINICAL TRIAL: NCT06948955
Title: Expanded Access to Bezuclastinib to be Coadministered With Sunitinib for Patients With Locally Advanced, Unresectable, or Metastatic Gastrointestinal Stromal Tumors
Brief Title: Expanded Access to Bezuclastinib to be Coadministered With Sunitinib for Patients With Gastrointestinal Stromal Tumors
Status: Available | Type: Expanded Access
Sponsor: Cogent Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CGT9486-EAP-002
Record Dates: First submitted 2025-03-31; First posted 2025-04-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Gastrointestinal Neoplasms, Gastrointestinal Stromal Tumors
Keywords: Solid Tumors; Sunitinib; Bezuclastinib; Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Neoplasms; Gastrointestinal Stromal Tumors | interventions — Sunitinib

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Bezuclastinib — Drug: Bezuclastinib
Drug: Sunitinib — Drug: Sunitinib (locally sourced)

SUMMARY:
The purpose of this expanded access program (EAP) is to provide investigational bezuclastinib so that it can be coadministered with sunitinib to patients with a diagnosis of gastrointestinal stromal tumors (GIST) with no comparable or satisfactory alternative therapy options. The combination of bezuclastinib and sunitinib provides broad inhibition of all primary and secondary KIT mutations that commonly occur in GIST.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent and commit to recommended EAP assessments.
* ≥18 years of age.
* Able to swallow tablets.
* Histologically confirmed locally advanced, metastatic, and/or unresectable GIST.
* Intolerant to imatinib or received prior imatinib therapy for treatment of advanced, metastatic, and/or unresectable GIST that resulted in disease progression.
* Meet clinically acceptable local laboratory results.

Exclusion Criteria:

* Patients who are eligible for and capable of participating in and/or enrolled in an on-going bezuclastinib clinical trial.
* Prior or known intolerance to sunitinib.
* Patients who have previously participated in a bezuclastinib clinical trial.
* Patients with persistent > Grade 2 toxicities from prior therapy.
* Known PDGFR driving mutations or known SDH deficiency.
* Pregnant or currently breastfeeding.

Other protocol-defined criteria apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Rachael Easton, MD, PhD, Study Director — Cogent Biosciences, Inc.
Locations (8):
- United States (8):
  - UCLA Department of Medicine- Hematology/Oncology, Los Angeles, California
  - Orlando Health, Orlando, Florida
  - The University of Chicago Medical Center, Chicago, Illinois
  - Dana Farber Cancer Institute (DFCI), Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - MD Anderson Cancer Center, Houston, Texas